CLINICAL TRIAL: NCT05180565
Title: Safe Anastomosis Feasibility Study: a Study to Investigate the Efficacy, Mechanism of Action and Safety of the Colovac+ Colorectal Anastomosis Protection Device
Brief Title: Safe Anastomosis Feasibility Study
Acronym: SAFE2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SafeHeal Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFE2019
Record Dates: First submitted 2021-10-26; First posted 2022-01-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Anastomosis
Keywords: anastomosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Colovac (Experimental): Patients receive Colovac device during colorectal surgery
  Interventions: Device: Colovac

INTERVENTIONS:
Device: Colovac — A removable, temporary intraluminal bypass device designed to safely postpone the creation of a protective stoma until 10 days after surgery for only patients who need it (do not have a healed anastomosis)

SUMMARY:
A clinical trial to assess the efficacy, mechanism of action and safety of the Colovac+ Colorectal Anastomosis Protection Device in providing temporary protection of the anastomosis in subjects undergoing lower anterior resection for colorectal cancer

DETAILED DESCRIPTION:
A primary diverting stoma is widely used by surgeons in order to bypass the low rectal anastomosis and reduce morbidity associated with anastomotic leaks. Typically, a stoma is created for all high-risk patients which means that many patients are exposed to potentially serious complications associated with the stoma itself without any clinical benefit.

Colovac+ is a local, temporary, minimally invasive bypass device that provides protection of the anastomosis and safely postpones stoma creation for 10 days after surgery. By postponing stoma creation for 10 days, Colovac is designed to avoid stoma creation in all patients except those patients whose anastomoses have not healed by 10 days after surgery, allowing the others to return to normal activity more quickly and safely.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older)
* Eligible to undergo open or minimally invasive sphincter-sparing low anterior resection with planned diverting loop ileostomy for malignancy, based on multidisciplinary team recommendations.
* Willingness to comply with Clinical Investigation Plan-specific treatment and study visits and to sign a written Informed Consent Form

Exclusion Criteria:

- Preoperatively :

1. Patient with inflammatory bowel disease
2. Known allergy to nickel or other components of the Colovac+ kit
3. Pregnant or nursing female subject
4. Concomitant major surgical procedure in combination with Colorectal resection (i.e. hepatectomy)
5. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation, impair the ability of the participant to undergo Clinical Investigation Plan described procedures or interfere with the interpretation of study results. including, but not limited to:

   1. COVID-19 positive (active infection) based on test within 72 hours prior to surgery
   2. Metastatic disease - unless previously treated with chemotherapy and resection, and the benefit of exposure to the Colovac device is greater than the risk 1
   3. Immunodeficiency (CD4+ count < 500 CU MM)
   4. Systemic steroid therapy within the past 6 months
   5. Systemic infection at the time of surgery or requiring systemic antimicrobial therapy up to 1 week before surgery
   6. Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
   7. Diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, intraabdominal infection, ischemic bowel, carcinomatosis
   8. Fecal incontinence, involvement of sphincter by the neoplastic disease or evidence of extensive local disease in the pelvis seen on pre-operative imaging
   9. Severe Malnutrition defined as 10% weight loss within 3 months prior to enrollment.
6. The subject is currently participating in another investigational drug or device study

   * Intraoperatively :
7. Anastomosis placement at more than 10cm from anal margin
8. Occurrence of any of the following during the colorectal surgery:

   1. Blood loss (>750 cc)
   2. Blood transfusion
   3. Any new sign of ischemia
   4. Positive air leak test - requiring re intervention on the anastomosis
   5. Inadequate bowel preparation
   6. Other intra-operative risks that preclude the subject from undergoing the procedure with the investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
To measure the incidence of serious adverse events related to using the device | 3 months
  The primary endpoint will be a measurement of SAEs probably related or causaly related to the use of the investigational device, to the index surgery in this clinical trial.

SECONDARY OUTCOMES:
To measure the number of participants with evidence of absence of feces between the sheath and the colonic wall before device retrieval | 10 days
  Rate of patients with evidence of absence of feces between the sheath and the colonic wall before device retrieval at 10 days:
To measure the rate of ostomy avoidance | 3 months
  To measure the number of participants where ostomy was avoided
To evaluate the occurrence of clinical anastomotic leakage | 3 months
To measure on a scale of 1 to 5 rated by the surgeon the ease of device introduction, positioning and endoscopic retrieval | 10 days
  * Ease of device introduction and positioning will be rated by the surgeon on a scale from 1 to 5 (1 being very easy and 5 being impossible)
  * Ease of endoscopic retrieval of the device will be rated by the endoscopist on a scale from 1 to 5 (1 being very easy and 5 being impossible)
To evaluate the clinically significant migration rate | 10 days
To evaluate the integrity above the anchoring site during the device retrieval using endoscopy. | 10 days
  Mucosal appearance above the anchoring site will be evaluated endoscopically during device retrieval and classified as Normal/Inflamed, Bleeding, Ulcerated, Perforated.
To evaluate the integrity of the anchoring site during the device retrieval using endoscopy. | 10 days
  Mucosal appearance at the anchoring site will be evaluated endoscopically during device retrieval and classified as Normal/Inflamed, Bleeding, Ulcerated, Perforated.
To evaluate the integrity of the anastomosis before the device retrieval using fluoroscopy | 10 days
  Fluoroscopy with injection of contrast between the colonic wall and the sheath will be performed prior to retrieval of the Colovac+ Device in order to check for anastomotic integrity before device retrieval.
  Outcome is measured with presence/absence of any contrast liquid leak through the anastomosis prior to device retrieval.
To evaluate the integrity of the anastomosis after the device retrieval using fluoroscopy | 10 days
  Fluoroscopy with injection of contrast per rectum will be performed immediately after retrieval of the Colovac+ Device in order to check for anastomotic integrity following device retrieval.
  Outcome is measured with presence/absence of any contrast liquid leak through the anastomosis after device retrieval.
To measure the average procedure time | 1 day
To measure the patient tolerability of the device using a patient questionnaire | 10 days
  Responses to a patient questionnaire on device acceptance, on the device handling and comfort, and on preference compared to an ostomy - utilizing the NIH's (National Institute of Health) PROMIS (Patient-Reported Outcomes Measurement Information System) health measurement questionnaires to assess parameters like pain, bowel incontinence, constipation, diarrhea, or anxiety and social isolation, on a scale from 1 to 10 (1 being absence of difficulty and 10 being severe problems).

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Lefevre, Principal Investigator — Hôpital Saint Antoine Paris
Locations (7):
- Belgium (2):
  - UZA, Antwerp
  - Centre Hospitalier Universitaire St Pierre, Brussels
- France (5):
  - CHU Lille, Lille
  - ICM Montpellier, Montpellier
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine Paris, Paris
  - CHRU Strasbourg, Strasbourg

REFERENCES:
- [Derived] De Hous N, D'Urso A, Cadiere GB, Cadiere B, Rouanet P, Komen N, Lefevre JH. Evaluation of the SafeHeal Colovac+ anastomosis protection device after low anterior resection for rectal cancer: the safe anastomosis feasibility evaluation (SAFE) 2019 trial. Surg Endosc. 2023 Sep;37(9):7385-7392. doi: 10.1007/s00464-023-10272-x. Epub 2023 Jul 18. PMID 37464064